CLINICAL TRIAL: NCT05532488
Title: The Inulin Effect on Burn-induced Insulin Resistance: a Randomized, Double-blind Placebo-controlled Pilot Trial
Brief Title: Inulin in Burn-induced Insulin Resistance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Marko Stojanovic, Assistant professor, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MicroModifiER
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Burn Injury; Insulin Resistance; Post Burn Insulin Resistance
MeSH Terms: conditions — Burns; Insulin Resistance | interventions — Inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inulin 20 mg (Experimental): Inulin 20 mg administrated orally q24h
  Interventions: Dietary Supplement: Inulin 20 mg
- Placebo (Placebo Comparator): Matching placebo q24h
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Inulin 20 mg — Inulin can increase gut Bifidobacterium count. Bifidobacterium has beneficial effects on the metabolic profile and insulin resistance biomarkers.
  Arms: Inulin 20 mg
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
In this clinical trial, investigators will test the effects of dietary supplement inulin, on the reduction of insulin resistance developed as a result of burn injuryy.

DETAILED DESCRIPTION:
As a consequence of burn injury, an exaggerated inflammatory response is developing in parallel with metabolic changes, which led to the development of hyperglycemia and insulin resistance. The post burn-injury insulin resistance is different in comparison to other trauma-induced insulin resistance. The main difference is the length. More precisely postburn-injury insulin resistance lasts longer than insulin resistance developed after other traumas. Insulin resistance can persist for years after the burn heals.

Inulin is a heterogeneous mixture of fructose polymers that are widely distributed in nature as storage of carbohydrates in plants. This mixture of fructose has nutritional value, but also affects general health, reducing the risk of developing various diseases. Inulin prevents gastrointestinal complications such as constipation, increases the resorption of minerals from the gastrointestinal tract, stimulates the immune system, and functions as a prebiotic, but can also affect insulin resistance in patients with metabolic syndrome.

The hypothesis: The everyday inulin can affect postburn-injury insulin resistance.

To investigate the effect of inulin on patients with postburn-injury insulin resistance a prospective, double-blind, randomized, and placebo-controlled clinical trial will be performed. This initial trial is a pilot trial. The pilot trial will be performed to assess the safety of treatment or interventions and recruitment potentials, examine the randomization and blinding process, increase the researchers' experience with the study methods and interventions, and provide estimates for sample size calculation for the main study.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent and willingness in study participation
* The age of the respondent greater than or equal to 18 years at the time of signing the informed consent
* Burns requiring in-hospital treatment
* insulin resistance detected on the fifth day of admission to the hospital

Exclusion Criteria:

* Documented pre-existing insulin resistance
* PCOS
* BMI ≥ 30 kg/m2
* Pregnancy
* Diabetes type 1
* Diabetes type 2
* Metabolic syndrome
* Use of drugs that can affect insulin resistance
* Weight loss greater than 10% in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Changes in insulin resistance measured by HOMA-IR | Baseline and end of the study (6week)
  Changes in insulin resistance in placebo and experimental group measured by HOMA-IR
Change in fasting plasma glucose level | Baseline and end of the study (6week)
  Changes in fasting plasma glucose in placebo and experimental group
Change in plasma insulin level | Baseline and end of the study (6week)
  Change in plasma insulin levelin placebo and experimental group
Changes in insulin resistance measured by QUICKI | Baseline and end of the study (6week)
  Changes in insulin resistance in placebo and experimental group measured by QUICKI
Changes in HbA1c level | Baseline and end of the study (6week)
  Changes in HbA1c level in placebo and experimental group

SECONDARY OUTCOMES:
Survival | 6 weeks
  The survival of patient in placebo and experimental group
Burn wound changes | 6 weeks
  The change in diameter, tissue type and contraction of wound in placebo and experimental group
Development of local and systemic infection | 6 weeks
  The developement of local and systhemic infection in placebo and experimental group

CONTACTS AND LOCATIONS:
Overall Officials: Marko A Stojanović, MD, PhD, Principal Investigator — University of Belgrade
Locations (1):
- Faculty of Medicine; Clinical Center of Serbia, Clinic for Burns, Plastic and Reconstructive Surgery, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be published before the beginning of the study. All of the other necessary information regarding the study will be available at Zenodo repository before publishing the data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The date of interest will be available at the beginning of study and at least three years after the termination of the study
Access Criteria: On demanded